CLINICAL TRIAL: NCT01639209
Title: A Randomised Controlled Trial Comparing Pneumatic Retinopexy Versus Vitrectomy for the Management of Primary Retinal Detachment; Anatomical Success, Functional Success and Impact on Patient Quality of Life
Brief Title: Pneumatic Retinopexy Versus Vitrectomy for Retinal Detachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB #12-031
Record Dates: First submitted 2012-07-09; First posted 2012-07-12 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: Retinal detachment; Pneumatic retinopexy; Vitrectomy
MeSH Terms: conditions — Retinal Detachment | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitrectomy (Experimental)
  Interventions: Procedure: Vitrectomy
- Pneumatic retinopexy (Experimental)
  Interventions: Procedure: Pneumatic retinopexy

INTERVENTIONS:
Procedure: Vitrectomy — Pars plana vitrectomy plus laser/cryotherapy
  Arms: Vitrectomy
Procedure: Pneumatic retinopexy — Pneumatic retinopexy plus laser/cryotherapy
  Arms: Pneumatic retinopexy

SUMMARY:
The purpose of this research study is to compare the outcomes of pneumatic retinopexy with the outcomes of vitrectomy (with or without scleral buckle) for the management of retinal detachment, in terms of anatomical success, functional success and impact on patient quality of life.

DETAILED DESCRIPTION:
Rhegmatogenous retinal detachment (RRD)is an acute, sight threatening condition, with an incidence of approximately 10 per 100,000 population. Both of the treatments under investigation are widely used and accepted by vitreoretinal surgeons, but randomised, prospective comparison of the two techniques has not been reported in the scientific literature to date. Currently, the management decisions surrounding primary retinal detachment are grounded on a weak evidence base. The findings of this study will allow vitreoretinal surgeons and their patients to select the most appropriate intervention for that individual, in an informed and holistic manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with acute rhegmatogenous retinal detachment
* Single retinal break OR group of breaks no larger than one clock hour (30°)
* All break/s in detached retina between 8-4 o'clock
* No significant proliferative vitreoretinopathy

Exclusion Criteria:

* Inferior breaks in detached retina
* Inability to read English language
* Age < 18 years
* Mental incapacity
* Previous vitrectomy (index eye)
* Previous retinal detachment (index eye)
* Inability to maintain the post-operative posturing
* Inability to carry out detailed examination of peripheral retina due to media opacity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 12 months post intervention

SECONDARY OUTCOMES:
Visual acuity | 1 week, 1 month, 3 months and 6 months post intervention
Subjective visual function | 3, 6 and 12 months post intervention
  Questionnaire
Anatomical success (complete retinal re-attachment) | 3, 6 and 12 months post intervention
Subjective health related quality of life | Baseline and 1 month post intervention
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev H Muni, FRCSC, Principal Investigator — St. Michael's Hospital (Toronto, Canada); Roxane J Hillier, FRCOphth, Principal Investigator — St. Michael's Hospital (Toronto, Canada)
Locations (1):
- Department of Ophthalmology, St Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Bansal A, Lee WW, Sarraf D, Sadda SR, Berger AR, Wong DT, Kertes PJ, Kohly RP, Hillier RJ, Muni RH. Persistent subfoveal fluid in pneumatic retinopexy versus pars plana vitrectomy for rhegmatogenous retinal detachment: posthoc analysis of the PIVOT randomised trial. Br J Ophthalmol. 2023 Nov;107(11):1693-1697. doi: 10.1136/bjo-2021-320981. Epub 2022 Aug 11. PMID 35953261
- [Derived] Muni RH, Felfeli T, Sadda SR, Juncal VR, Francisconi CLM, Nittala MG, Lindenberg S, Gunnemann F, Berger AR, Wong DT, Altomare F, Giavedoni LR, Kohly RP, Kertes PJ, Sarraf D, Hillier RJ. Postoperative Photoreceptor Integrity Following Pneumatic Retinopexy vs Pars Plana Vitrectomy for Retinal Detachment Repair: A Post Hoc Optical Coherence Tomography Analysis From the Pneumatic Retinopexy Versus Vitrectomy for the Management of Primary Rhegmatogenous Retinal Detachment Outcomes Randomized Trial. JAMA Ophthalmol. 2021 Jun 1;139(6):620-627. doi: 10.1001/jamaophthalmol.2021.0803. PMID 33885738
- [Derived] Muni RH, Francisconi CLM, Felfeli T, Mak MYK, Berger AR, Wong DT, Altomare F, Giavedoni LR, Kohly RP, Kertes PJ, Figueiredo N, Zuo F, Thorpe KE, Hillier RJ. Vision-Related Functioning in Patients Undergoing Pneumatic Retinopexy vs Vitrectomy for Primary Rhegmatogenous Retinal Detachment: A Post Hoc Exploratory Analysis of the PIVOT Randomized Clinical Trial. JAMA Ophthalmol. 2020 Aug 1;138(8):826-833. doi: 10.1001/jamaophthalmol.2020.2007. PMID 32556156